CLINICAL TRIAL: NCT01774734
Title: Effect of Combined Neck Strength Exerciser Plus Physiotherapy in Treatment of Patients With Chronic Neck Pain
Brief Title: Effect of Combined Neck Strength Exerciser Plus Physiotherapy to Treatment Chronic Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20110605R
Record Dates: First submitted 2012-07-23; First posted 2013-01-24 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Cervicalgia
Keywords: Chronic neck pain; Neck strength exerciser; Biofeedback; Physiotherapy; Strengthening exercise; Randomized trials
MeSH Terms: conditions — Neck Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- neck strength exerciser (NSE) group (Experimental): Traditional physiotherapy 30 minutes per session for three times weekly + home-based NSE training 20 minutes daily
  Interventions: Other: Physical therapy; Device: Neck Strength Exerciser (NSE)
- Physical therapy group (Placebo Comparator): Traditional physiotherapy 30 minutes per session for three times weekly + home-based general neck exercise 20 minutes daily
  Interventions: Other: Physical therapy

INTERVENTIONS:
Other: Physical therapy — Physical therapy
  * Provided by 2 experienced physiotherapist
  * Applied to every patients 3 times weekly
Device: Neck Strength Exerciser (NSE) — * Neck strength exerciser use 10-20 minutes daily at home
  * Plus traditional physical therapy three times weekly provided by two experienced physical therapist
  Arms: neck strength exerciser (NSE) group

SUMMARY:
1. Chronic neck pain is common in general population.

   * High health care source expenditure
   * Multiple therapeutic approaches available with limited evidence
   * Previous studies showed active strengthening exercise improved pain (VAS) and functional performance (NDI)
   * Muscle strengthening exercise with biofeedback technique showed more long-lasting effect in patients with chronic neck pain
2. The investigators hypothesize that daily use of the neck strength exerciser (NSE), combined biofeedback technique with muscle strengthening exercise posture adjustment, in addition to traditional physiotherapy, could have more long-lasting and prominent effect on pain and functional improvement in patients with chronic neck pain.

DETAILED DESCRIPTION:
1. A randomized single-blinded trial to compare the effect of combined home-based NSE with physiotherapy could be more effective to treat people with chronic neck pain

* The NSE is a simple equipment that is easy to learn and safe to apply as home-based program
* The NSE will apply to the patients in the NSE group for 6 weeks, and we will compare the target variables to see if it brings better improvement by correction of maladaptive habitual posture and daily postural muscle exercise

ELIGIBILITY:
Inclusion Criteria:

* Adult, ≧20 yr.
* Constantly or frequently occurring neck pain for more than 3 months in the last 1 year.
* Motivated and willing to participate in rehabilitation therapy
* Sign written informed consent.

Exclusion Criteria:

* Neck or shoulder surgery.
* Clinical evidence of cervical radiculopathy or myelopathy.
* History of disk disease, degenerative joint disease, fracture, or dislocation in the cervical vertebrae.
* Severe pathological change in the cervical vertebrae, including inflammatory rheumatic disease and tumor.
* History of poor diet, hypothyroidism, or other severe systemic disorders.
* Cognitive deficit and severe psychiatric illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Visual analog scale (VAS) at three-month interval | day 0; day 42; 12 weeks
  a 10-point horizontal line with 0 represented the expressions "no pain at all, and 10 represented "the most intense pain imaginable"

SECONDARY OUTCOMES:
Cervical active ROM | day 0; day 42; 12 weeks
  including flexion, extension, side bending, and rotation was measured a special cervical goniometer (CROM)
Patient global assessment (PGA) | day 0; day 42; 12 weeks
  The PGA questions will ask: "How has the neck pain been at the present time?" and will be scored on a Likert scale(very good＝1; good＝2; fair＝3; poor＝4; very poor＝5)
Neck Disability Index (NDI) | day 0; day 42; 12 weeks
  The NDI was developed and validated by Vernon et al to measure neck pain and disability.[5] It is a 10-item self report instrument that evaluates perceived disability in 10 areas: pain intensity, self care, lifting, reading, headache, attention, working, driving, sleep and leisure activity. By using a 6-point Likert scale (1= no limitation; 6= severe limitation), the total maximal score was calculated. (appendix)
Effect of the intervention on the neck pain | day 42; 12 weeks
  on a 6-point scale: 1 indicating more pain, and 6 indicating for completely relief from pain
Amount of sick leave | day 42; 12 weeks
Amount of analgesics | day 42; 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D., Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan